CLINICAL TRIAL: NCT01026922
Title: Use of an Ambulatory Capsule to Characterize Gastrointestinal Pressure Patterns in Children
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: The SmartPill Corporation (Industry)
Responsible Party: Principal Investigator, Carlo Di Lorenzo, Division Chief, Nationwide Children's Hospital
Other Study IDs: NCHSmartPill-01
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Upper Gastrointestinal Motility Disorders
Keywords: antroduodenal manometry; gastric dysmotility; intestinal dysmotility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SmartPill Participants: It is a single-center study, children aged 8-17 years with severe upper GI symptoms (ie, nausea, vomiting, retching, abdominal pain) referred for antroduodenal manometry (ADM) studies underwent a wireless motility capsule (smartpill) test. The scintigraphic gastric emptying study was done when clinically indicated either at the time of the ADM or at a different time within 1 year of the wireless motility capsule test. In summary, we studied symptomatic adolescents using scintigraphic gastric emptying studies, ADM, and the wireless motility capsule test, with the goal of identifying the diagnostic yield of each test and exploring how they compare in detecting motor abnormalities in the GI tract.

SUMMARY:
This study will test a new medical device called the SmartPill GI Monitoring System, which is now used to diagnose gastric motility disorders in adults, in children. The study will compare the SmartPill capsule findings to antroduodenal manometry (ADM), which is a standard procedure currently used for the evaluation of gastric and duodenal motility in children. The ADM studies will be done for clinical purposes and only if recommended by the patient's gastroenterologist. The research portion of the study is limited to the use of SmartPill.

DETAILED DESCRIPTION:
ADM is a standard procedures used in children, but it has some limitations and disadvantages. Manometry studies involve placing catheters in the nose and are often poorly tolerated by children. Also, placement of the catheter requires sedation or anesthesia, the manometry test lasts several hours and involves ingestion of a meal which many children find difficult when having a catheter in their nose. The reason we are conducting this study is because we would like to find a new, less invasive, equally informative test for understanding gastrointestinal motility.

The SmartPill GI Monitoring System uses a capsule, about the size of a large vitamin or PillCam capsule, which is swallowed and passed through the stool. While in the GI tract, the capsule measures the acidity (pH) and pressures, and these measurements are used to determine how long it takes for food to leave the stomach. Pressure and pH information are sent by the capsule to a receiver that the patient will either wear on the belt or keep within 2 feet. The receiver stores data collected about the pH, temperature, and pressure inside the GI tract. The SmartPill GI Monitoring System has already been approved by the Food and Drug Administration (FDA) for use in adults but not in children.

ELIGIBILITY:
Inclusion Criteria:

* Children older than 10 years of age referred to our Motility Center to receive AD manometry studies will be offered participation to the study
* The patients will have to be able to swallow the SmartPill capsule
* The patients will need to have no evidence of strictures or narrowing

Exclusion Criteria:

* Inability to swallow the capsule
* Patients on TPN because of inability to tolerate enteral feedings (high likelihood of not emptying the capsule from the stomach)
* Children with evidence of strictures
* Children with history of esophageal or gastric surgeries, such as TE fistula, fundoplication, or gastrojejunostomy
* Children with a history of gastric bezoars
* Allergies to components of the test meal including eggs, bread, and jam
* Patients with history of inflammatory bowel disease

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients coming to clinic for concerns of gastric or small bowel dysmotility
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Determine if a patient's gastric and duodenal motility is considered normal or abnormal, if their motility disorder considered as neuropathic (normal amplitude of contractions) or myopathic (low amplitude or absent contractions) based on ADM vs SmartPill | SmartPill use will be within 180 days of ADM
  Determine if a patient's gastric and duodenal motility is considered normal or abnormal, if their motility disorder considered as neuropathic (normal amplitude of contractions) or myopathic (low amplitude or absent contractions) based on ADM vs SmartPill. The goal is to identify the diagnostic yield of each test and exploring how they compare in detecting motor abnormalities in the GI tract.

SECONDARY OUTCOMES:
The patient's tolerance using the Smartpill | The day the patient returns the SmartPill recording device
  Assess the tolerability and safety of the wireless motility capsule test.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Di Lorenzo, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Center for Digestive Disorders at Nationwide Childrens Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuo B, McCallum RW, Koch KL, Sitrin MD, Wo JM, Chey WD, Hasler WL, Lackner JM, Katz LA, Semler JR, Wilding GE, Parkman HP. Comparison of gastric emptying of a nondigestible capsule to a radio-labelled meal in healthy and gastroparetic subjects. Aliment Pharmacol Ther. 2008 Jan 15;27(2):186-96. doi: 10.1111/j.1365-2036.2007.03564.x. Epub 2007 Oct 28. PMID 17973643
- [Background] Cassilly D, Kantor S, Knight LC, Maurer AH, Fisher RS, Semler J, Parkman HP. Gastric emptying of a non-digestible solid: assessment with simultaneous SmartPill pH and pressure capsule, antroduodenal manometry, gastric emptying scintigraphy. Neurogastroenterol Motil. 2008 Apr;20(4):311-9. doi: 10.1111/j.1365-2982.2007.01061.x. Epub 2008 Jan 13. PMID 18194154
- [Background] Rao SS, Kuo B, McCallum RW, Chey WD, DiBaise JK, Hasler WL, Koch KL, Lackner JM, Miller C, Saad R, Semler JR, Sitrin MD, Wilding GE, Parkman HP. Investigation of colonic and whole-gut transit with wireless motility capsule and radiopaque markers in constipation. Clin Gastroenterol Hepatol. 2009 May;7(5):537-44. doi: 10.1016/j.cgh.2009.01.017. PMID 19418602